CLINICAL TRIAL: NCT04780698
Title: DCI COVID-19 Surveillance Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 27042
Record Dates: First submitted 2021-02-12; First posted 2021-03-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Cohort (Experimental)
  Interventions: Diagnostic Test: SARS-CoV-2 RT-PCR Assay for Detection of COVID-19 Infection

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 RT-PCR Assay for Detection of COVID-19 Infection — COVID-19 infection and antibody testing
  Other Names: Beckman Coulter Access SARS-CoV-2 IgG Antibody Test

SUMMARY:
This is a prospective longitudinal census study conducted at a single center (DCI Inc., Henry Avenue, Philadelphia). The purpose of this study is to gain information about COVID-19 infection and antibody response in an in-center dialysis population. The investigators hypothesize that screening and surveillance for COVID-19 positive test (viral infection) and antibodies response to infection (potential immunity) in a dialysis center population within a high-prevalence region can provide foundational information to guide approaches toward prevention of COVID-19 related illness in a susceptible population. Participants will be given a questionnaire initially and monthly over the study period to find out whether they have had COVID-19 infection, hospitalization, or symptoms. A nasopharyngeal swab test for COVID-19 infection and a blood sample for COVID-19 antibody will be collected monthly for the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive in-center chronic dialysis (>3 months) at DCI Henry Avenue
* Patients who are able to consent for study

Exclusion Criteria:

* Patients receiving transient hemodialysis at DCI or receiving hemodialysis for Acute Renal Failure
* Patients who are unable to consent
* Patients who are receiving other forms of dialysis therapy (e.g. home hemodialysis, peritoneal dialysis)
* Patients whose life expectancy is <12 months
* Patients who are planning to leave the dialysis center within 12 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 infection in the cohort | monthly through study completion (average of 18 months)
  COVID-19 infection assessed using the Hologic Aptima SARS-CoV-2 Assay and/or the Luminex NxTAG SARS-CoV-2 Extended Panel
Link the presence of COVID-19 infection to COVID-19 antibody formation (seroconversion) from qualitative testing | monthly through study completion (average of 18 months)
  Antibody formation assessed using the Beckman Coulter Access SARS-CoV-2 IgG Antibody Test
Incidence of COVID-19 reinfection | monthly through study completion (average of 18 months)
  COVID-19 infection assessed using the Hologic Aptima SARS-CoV-2 Assay and/or the Luminex NxTAG SARS-CoV-2 Extended Panel
Presence of antibodies in cases of reinfection | monthly through study completion (average of 18 months)
  Antibody formation assessed using the Beckman Coulter Access SARS-CoV-2 IgG Antibody Test

CONTACTS AND LOCATIONS:
Overall Officials: Avrum Gillespie, MD, Principal Investigator — Temple University
Locations (1):
- Dialysis Clinic, Inc., Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No